CLINICAL TRIAL: NCT02468076
Title: Investigation of the Effect of Intraductal Radiofrequency Ablation in Inoperable Biliopancreatic Tumors Complicated With Obstructive Jaundice
Brief Title: Radiofrequency Ablation for Biliopancreatic Malignancy
Acronym: IGNITE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGNITE-1
Record Dates: First submitted 2015-01-05; First posted 2015-06-10 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2014-11

CONDITIONS: Pancreas Cancer; Cholangiocarcinoma; Obstructive Jaundice
Keywords: ERCP; radiofrequency ablation; obstructive jaundice
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Jaundice, Obstructive | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiofrequency ablation (StarMed) (Experimental): Radiofrequency ablation catheter
  Interventions: Device: Radiofrequency ablation (StarMed)

INTERVENTIONS:
Device: Radiofrequency ablation (StarMed) — Radiofrequency ablation into bile duct

SUMMARY:
This phase-2 study aims to evaluate feasibility, safety and efficacy of thermal ablation of biliary obstructive malignancies by means of radiofrequency ablation (RFA, ELRA, StarMed) during endoscopic retrograde cholangio-pancreaticography (ERCP) with primary intent to obtain palliative biliary drainage via stenting

DETAILED DESCRIPTION:
INTRODUCTION

Biliary obstruction is the most relevant factor for survival and quality of life in patients suffering from primary bile duct malignancies or pancreatic head carcinoma. Due to their insidious course, these cancers are often diagnosed at an advanced stage. Thus, therapy is frequently restricted to palliative management. Within this setting, the prevention/treatment of biliary complications such as jaundice, cholangitis, or sepsis is one of the key therapeutic factors to extend survival and maintain quality of life (1-3). Endoscopic stenting of the biliary tract is now generally accepted as the primary approach to reestablish sufficient biliary drainage, provided approximately 50% of the liver parenchyma is drained (4). As the tumor grows, unfortunately, it often occurs that jaundice reappears despite primary stenting. Most oftenly this relates to unbridled tumor expansion leading to either stent-dysfunction by tumor ingrowth (through the mesh in case of metallic stenting of or via clogging of plastic stents) or either to extension in more proximal bile ducts/branches shutting of sufficient/adequate biliary drainage.

Given the context of incurable disease, a minimally-invasive strategy that could reduce the tumor burden in addition to stenting might be considered beneficial in terms of longer sustained bile duct drainage, and as such improve quality of life, more efficiently administered and better tolerated courses chemotherapy and delayed disease progression.

An example of such a potential minimal invasive strategy is RadioFrequency Ablation (RFA). It involves a modified electrocautery technique that has emerged among the many choices for local, minimally invasive tissue ablation. It has proven effective, versatile, and relatively inexpensive. RFA has been used for years in the treatment of cardiac dysrhythmias from aberrant conduction pathways, osteoid osteoma, prostate hypertrophy, and chronic pain (5-8). Recent clinical applications include tumor ablation in the liver (9-11), kidney (12,13) adrenal gland (14,15), bone (16), lung (17), and breast (18) as well as soft tissue debulking and pain palliation (19).

In the context of gastro-intestinal endoscopy, RFA has taken its place in the reduction of neoplastic progression of Barrett esophagus over 3 years of follow-up (20).

With regard to biliopancreatic endoscopy and oncology in particular, this approach has only recently been introduced. A primary experience using an alternative endoscopically applicable RFA-system for bile duct lesions, has shown to be feasible and safe ex vivo in resected fresh pig livers and in an open-label pilot study involving 22 patients with malignant biliary obstruction (21,22). Similar results have been obtained in animal testing for the ELRA-system (StarMed, Taewoong Medical, Seoul, Korea).

The presumed theoretical advantage of the current system (ELRA system, StarMed, Taewoong Medical, Seoul, Korea) is the capacity to better control the locally applied temperature at all times and to maintain temperature continuous, as such preventing tissue adjacent to an active tip from carbonization during the procedure. Additionally the 4-ring appliance of thermal ablation allows a better thermal spreading and therefore appliance of ablation

STUDY OBJECTIVE & DESIGN

This project involves a single center investigator-driven prospective non-randomized non-controlled trial evaluating feasibility, safety and efficacy of thermal ablation of biliary obstructive malignancies by means of the ELRA RF during ERCP with primary intent to obtain palliative biliary drainage via stenting .

STUDY METHODOLOGY : POPULATION & INTERVENTION

ELIGIBLE PATIENT POPULATION

All patients with an inoperable biliopancreatic tumor with obstructive jaundice and therefore in need of biliary drainage via ERCP, eligible and consenting for inclusion (cfr infra), will be considered for entry in the study. This is a non-randomized non-controlled investigator-driven trial.

ENDOSCOPIC INTERVENTION

All procedures will be performed under general anesthesia, according to standard good clinical practice. After performing an endoscopic sphincterotomy with/without balloon dilatation of the stenosis (conventional approach) in preparation of stenting, a RFA catheter (ELRA, Taewoong, Seoul, Korea), suitable for endoscopic delivery into the biliary tree over a 0.035-inch guide wire, will be advanced up to the level of the malignant stenosis.

The "end of follow-up" is defined as the end of the follow-up period (designated at 3 months after index procedure) or failure of treatment or death.

The outcome parameters will be compared to those of a historically matched control group (i.e. stented without RFA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects with age above 18 years old
2. A confirmed diagnosis (endoscopic radiology, histology etc) of pancreatic or cholangiocarcinoma with obstructive jaundice considered inoperable according to multidisciplinary assessment
3. Willing and able to give written informed consent

Exclusion Criteria:

1. Refusal to consent or undergo ERCP
2. Less than 50% of liver parenchyma potentially drainable on pre-intervention imaging
3. Platelets < 40 x 109 mm3, an international normalized ratio (INR) > 1.5
4. Other concomitant disease or condition likely to significantly decrease life expectancy (e.g., moderate to severe congestive heart failure, severe COPD)
5. Portal vein thrombosis

18 patients to be included : Hilar cholangiocarcinoma : n=9 Distal cholangiocarcinoma/pancreatic cancer n=9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Feasibility (ratio of technically successful RFA-applications to all examinations in which RFA-use was intended) | 90 days after index procedure

SECONDARY OUTCOMES:
Efficacy measured by progression-free survival at 3 months upon standard follow-up imaging study and duration of stent patency (days) after the RFA-performed procedure | 90 days after index procedure
30-day-, 90-day and overall mortality | 90 days after index procedure
Number of days and reasons for hospitalizations during the study period | 90 day after index procedure
Quality of life (QuoL) by means of the EORTC QLQ-C15-PAL questionnaire after the procedure and at 30 and 90 days vs before | 90 days after index procedure
safety (number and type of adverse events) | 90 days after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Laleman Wim, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Brabant, Belgium

REFERENCES:
- [Derived] Laleman W, van der Merwe S, Verbeke L, Vanbeckevoort D, Aerts R, Prenen H, Van Cutsem E, Verslype C. A new intraductal radiofrequency ablation device for inoperable biliopancreatic tumors complicated by obstructive jaundice: the IGNITE-1 study. Endoscopy. 2017 Oct;49(10):977-982. doi: 10.1055/s-0043-113559. Epub 2017 Jul 21. PMID 28732391